CLINICAL TRIAL: NCT06407115
Title: Adapting and Implementing a Nurse Care Management Model to Care for Rural Patients With Chronic Pain
Acronym: AIM-CP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Sebastian Tong, Associate Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019595; 1UG3NR020930 (NIH); 4UH3NR020930-02 (NIH)
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
Keywords: chronic pain; behavioral health; rural health; telehealth; exercise
MeSH Terms: conditions — Chronic Pain; Motor Activity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Phase 1: Feasibility phase with a single intervention arm. Phase 2: RCT with two arms: the NCM model and treatment as usual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse Care Manager Arm (Experimental): In this feasibility pilot, all participants will be assigned to work with a care manager for 6 months and receive all components of the intervention. The care manager will meet with participants in virtual appointments every month to create a care plan and monitor progress. The program will also include: 6-10 sessions of Cognitive Behavioral Therapy (CBT) for chronic pain, which focuses on skills and strategies to empower participants to better manage their pain. Finally, the Care Manager will help counsel participants on physical exercise and refer patients to tele-EnhanceFitness, an online community program that allows users to access instructor-led group exercise classes from home.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Exercise Counseling and tele-EnhanceFitness; Other: Care Coordination; Other: Standard Clinical Practice Regimen
- Treatment as Usual (Active Comparator): In the Treatment as Usual arm, participants will continue receiving routine care from their primary care team. This may include referrals to specialists or allied health professionals, Given the heterogeneity among patients and between sites, it will be characterized in research assessments to allow for transparent reporting.
  Interventions: Other: Standard Clinical Practice Regimen

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — CBT in this study will consist of a series of 6-10, 30-45-minute sessions with the care manager. These 1-on-1 sessions will occur every week or every other week virtually. Content will be focus on addressing unhelpful thinking and small behavioral changes that may help participants better manage their pain.
  Arms: Nurse Care Manager Arm
Behavioral: Exercise Counseling and tele-EnhanceFitness — Participants will be counseling on physical exercise and encouraged enroll in instructor-led exercises classes for up to an hour, 3 days per week. These classes can be accessed from home. Data plans and tablets are available to aid participants that need them to gain access to the classes.
  Arms: Nurse Care Manager Arm
Other: Care Coordination — Care manager will meet with patient in virtual sessions once a month to create a care plan and monitor progress. Care manager will assess social determinants of health and link participants to resources in the community as appropriate. In addition, participants will take monthly assessments about pain and mood to help guide clinical decision making.
  Arms: Nurse Care Manager Arm
Other: Standard Clinical Practice Regimen — Routine clinical care provided by the primary care team. This may include, consultations, medications, and referrals.

SUMMARY:
Chronic pain affects over 20% U.S. adults and has debilitating effects on quality of life and physical and mental health. Individuals living in rural communities experience higher rates of chronic pain as well as poorer health outcomes due to pain. The 46 million Americans who live in rural areas frequently lack access to evidence-based, non-pharmacologic treatments for chronic pain. As such, a critical need exists to implement effective, comprehensive programs for pain management that include treatment options other than medications. Nurse care management (NCM) has been successfully used to enhance care for individuals with other long-term health issues. The study teams proposes to adapt, pilot, and implement a NCM model that includes care coordination, cognitive behavioral therapy (CBT), and referrals to a remotely delivered exercise program for rural patients with chronic pain.

DETAILED DESCRIPTION:
Care managers will provide care coordination to help patients address their health holistically and help link them key resources in the community. In addition, the care managers will be trained to deliver cognitive behavioral therapy (CBT) to address unhelpful thought patterns and behaviors around chronic pain and also facilitate patients' participation in physical exercise. One exercise option offered is EnhanceFitness (tele-EF), an evidence-based exercise program that can be accessed from home. The rationale is that both tele-EF and CBT have been independently shown to improve pain, functioning, and quality of life and that care managers could support patients in accessing and engaging in these services.

Phase 1 allowed the study team to prepare for a randomized controlled trial to test the adapted NCM model with rural patients who have chronic pain. Investigators assessed feasibility of implementing this intervention in rural serving health care systems using two practice-based research networks with substantial rural presence, the WWAMI (Washington, Wyoming, Alaska, Montana, and Idaho) region Practice and Research Network and Mecklenburg Area Partnership for Primary Care Research in North Carolina. In combination, recruitment in these two networks will allow the study team to reach ethnically diverse participants across broad rural geographies.

Phase 2 is the randomized controlled trial across multiple sites of the integrated NCM model to test whether it is effective in reducing pain interference.

ELIGIBILITY:
Inclusion Criteria:

* Current primary care patient with one care visit in the last year
* Experience pain for at least 3 months
* Live in a rural area
* Proficient in English
* A total score ≥ 12 on the 3-item Pain, Enjoyment, and General Activities scale

Exclusion Criteria:

* Pain is cancer-related
* Current treatment with chemotherapy and/or radiation therapy regardless of underlying diagnosis
* Scheduled surgical procedures in the next 6 months
* Has received skills training or education for pain management in the past 6 months
* Moderate or severe cognitive impairment (documented Alzheimer's or dementia diagnosis in EHR or score 12 or lower on the telephone Montreal Cognitive Assessment)
* On palliative care or living in a nursing home or inpatient treatment facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Pain Interference | Baseline, Post-intervention (6 months after baseline), 12-month follow-up
  The Pain, Enjoyment and General Activities scale is a validated 3-item, 0-10 rating scale that measures pain intensity and pain interference with enjoyment of life and general activity. The 3 items are averaged to get the mean score (out of 10). A higher score indicates more severe pain and pain-related interference with life and activities.

SECONDARY OUTCOMES:
Physical functioning | Baseline, Post-intervention (6 months after baseline), 12-month follow-up
  The Patient Reported Outcomes Measurement Information (PROMIS) pain interference short form (version 6b) measures changes in functionality. Scores range from 6-30 that are converted to T-scores with a range of 0-100. Higher scores indicate better physical functioning.
Pain catastrophizing | Baseline, Post-intervention (6 months after baseline), 12-month follow-up
  The Patient Reported Outcomes Measurement Information (PROMIS) 6-item pain catastrophizing scale indicates the degree to which respondents have thoughts and feelings when they are experiencing pain. Scores are computed on a scale of 0-24 with higher scores indicating more catastrophic thoughts.
Sleep Disturbance | Baseline, Post-intervention (6 months after baseline), 12-month follow-up
  The Patient Reported Outcomes Measurement Information (PROMIS) 6-item sleep disturbance short form (version 6a) represents how much difficulty respondents have with sleep. It is scored from 6 to 30 and then converted to T-scores 0-100 with higher scales indicating more sleep problems.
Depression | Baseline, Post-intervention (6 months after baseline), 12-month follow-up
  The Personal Health Questionnaire (8-item) measures depressions symptoms. Scores range from 0 to 24 with higher scores indicating more severe depression.
Anxiety | Baseline, Post-intervention (6 months after baseline), 12-month follow-up
  The General Anxiety Disorder (7-item) measures anxiety symptoms. Scores range from 0 to 21 with higher scores indicating more severe anxiety.
Unhealthy Substance Use | Baseline, Post-intervention (6 months after baseline), 12-month follow-up
  The Tobacco, Alcohol, Prescription Medication, and Other Substance Use tool is a 4-item screener that identifies unhealthy substance use. Sum scores are not calculated for the 4-item screener. Unhealthy use is any use for the questions about prescription medication and other drugs and monthly use or more for the questions about tobacco and alcohol.
Opioid Medication Exposure | Baseline, Post-intervention (6 months after baseline), 12-month follow-up
  Morphine Milligram Equivalents calculated by extracting prescription data from the electronic health record.
Health Service Utilization | Baseline, Post-intervention (6 months after baseline), 12-month follow-up
  Patient reported accounting of health services such as physical therapy, behavioral, primary care, urgent care, emergency room visits and referrals and appointments with specialists and/or allied health professionals (e.g., physical therapy, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Tong, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Atrium Health/Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All trial outcomes data will be shared according to HEAL Initiative standards in the NIMH Data Archive.